CLINICAL TRIAL: NCT06169462
Title: Comparison of Pericapsular Nerve Group (PENG) Block Alone Versus Combined With Suprainguinal Fascia Compartment Block (SIFCB) for Postoperative Analgesia and Quality of Recovery in Older Adult Patients With Hip Fractures
Brief Title: Comparison of Pericapsular Nerve Group Block With Suprainguinal Fascia Compartment Block in Hip Fractures
Status: Completed | Type: Observational
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 10-2023/17
Record Dates: First submitted 2023-11-21; First posted 2023-12-13 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Hip Fractures
Keywords: Anesthesia; Lower extremity; pericapsular nerve group block; suprainguinal fascia compartment block
MeSH Terms: conditions — Hip Fractures | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pericapsular nerve group (PENG) block: Patients who underwent PENG in Hip surgery under spinal anesthesia will be evaluated retrospectively in terms of opioid consumption and NRS scores.
  Interventions: Procedure: PENG block
- Suprainguinal fascia compartment block (SIFCB) + PENG: Patients who underwent PENG+SIFCB in Hip surgery under spinal anesthesia will be evaluated retrospectively in terms of opioid consumption and NRS scores.
  Interventions: Procedure: PENG block+ SIFCB

INTERVENTIONS:
Procedure: PENG block — Patients underwent ultrasound-guided PENG Block for older adult patients surgery for hip fracture. Patients who received opioids as a rescue analgesic during postoperative pain management on selected dates will be included in the study.
  Other Names: Drug
  Groups: Pericapsular nerve group (PENG) block
Procedure: PENG block+ SIFCB — Patients underwent ultrasound-guided PENG Block+ SIFCB for older adult patients surgery for hip fracture. Patients who received opioids as a rescue analgesic during postoperative pain management on selected dates will be included in the study.
  Other Names: Drug
  Groups: Suprainguinal fascia compartment block (SIFCB) + PENG

SUMMARY:
Ultrasound-guided Supra-inguinal Fascia Iliaca compartment Block (SIFCB) and Pericapsular Nerve Group Block (PENG) are increasingly being used for postoperative analgesia for hip surgery. The postoperative analgesic efficacy of SIFCB added to PENG block in elderly hip fracture patients will be evaluated. Postoperative opioid consumption and quality of recovery will also be evaluated.

DETAILED DESCRIPTION:
The study was conducted as a retrospective cohort feasibility design within a tertiary hospital. Patient records and electronic data systems were used to gather the required data for analysis. Before surgery, a carefully selected cohort of patients who underwent PENG block and PENG block added SIFCB were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Physical status according to American Society of Anesthesiologists (ASA ) I-III

Exclusion Criteria:

* Previous operation on the same hip
* Hepatic or renal insufficiency
* Patients undergoing general anesthesia
* Allergy or intolerance to one of the study medications
* BMI >40
* ASA IV

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Data of patients underwent hip surgery under spinal anesthesia between 31.01.2023 and 01.10.2023.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | Postoperative 48th hour
  If the patient's Numerical Rating Scale (NRS) score is equal to or above 4, tramadol 50 mg IV or oxycodone 5 mg orally every 4 hours will be administered as rescue analgesia.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) scores | Postoperative 48th hour
  Range 0-10, 0=no pain, 10=the worse pain ever
Quality of Recovery 15 Score | Postoperative day 1 and 1 month
  Quality of Recovery (QoR)-15 survey.Minimum value: 0, Maximum value: 150, higher scores mean better
Postoperative complications | 24 hours
  Presence of postoperative nausea, vomiting, pruritus, urinary retention, respiratory depression
Mobilization time | 24 hours
  Mobilization time

CONTACTS AND LOCATIONS:
Locations (1):
- Karaman Training and Research Hospital, Karaman, Karaman/Merkez, Turkey (Türkiye)